CLINICAL TRIAL: NCT07381647
Title: Clinical Observation of Facial Acupuncture for Insomnia Based on Zangfu Meridian Theory
Brief Title: Clinical Observation of Facial Acupuncture for Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pei Yuan (Other)
Responsible Party: Sponsor-Investigator, Pei Yuan, lecturer, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202510268122
Record Dates: First submitted 2026-01-07; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facial acupuncture treatment group (Experimental)
  Interventions: Procedure: facial acupuncture
- Facial scraping treatment group (Active Comparator)
  Interventions: Procedure: facial scraping

INTERVENTIONS:
Procedure: facial acupuncture — Acupuncture at specific points, each time leaving the needle for 30 minutes, twice a week, for four weeks.
  Arms: Facial acupuncture treatment group
Procedure: facial scraping — Scrape the specific areas of the face, each time for 15-20 minutes, twice a week, with an interval of at least 2, for 4 weeks continuously, a total of 8 times.
  Arms: Facial scraping treatment group

SUMMARY:
Insomnia is one of the most common mental disorders and has shown an upward trend in recent years. The commonly used western medicine treatment methods are easy produce drug-related adverse reactions, and there are problems such as the decline of efficacy and the production of drug dependence after long-term medication. Traditional Chinese medicine treatment of insomnia on syndrome differentiation. In this study, taking the common heart and spleen deficiency syndrome and liver depression transforming into fire syndrome as examples, based on the theory of zangfu andingluo, we explored the selection of acupoints for acupuncture treatment of insomnia and conducted clinical efficacy observation. Combined with the analysis of the changes of Pittsburgh Quality Index, Hamilton Anxiety Scale, Traditional Chinese Medicine Syndrome Efficacy Rating, Infrared Thermal Image Acquisition, Forehead Adhesive Sleep Recorder and other data, the acupuncture treatment of insomnia patients was expounded.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for insomnia in both Western and traditional Chinese medicine and the classification criteria for TCM syndrome differentiation;
* Between 16 and 30 years old (including 16 and 30 years old);
* No mental or language disorders;
* PQSI score ≥ 7;
* No hypnotic medication treatment within two weeks before the study;
* Patient informed consent, and voluntarily participate in this.

Exclusion Criteria:

* Those who do not meet the above inclusion criteria;
* Those with secondary insomnia caused by organic diseases, mental diseases etc.;
* Those who faint at acupuncture or refuse acupuncture;
* Those who have received any facial acupuncture or thread embedding within 3 months;
* Those who have received radiofrequency or laser wrinkle removal treatment within half a year;
* Those who have received facial tissue filler injection and A-type botulinum toxin injection and other long-term facial rejuvenation treatment within one year;
* Pregnant or lactating, those preparing for pregnancy during the treatment process;
* Those who work night shifts for a long time, with irregular work and rest;
* Those withocrine function, immune function diseases, and those with severe primary diseases of the heart, brain, liver, kidney and hematopoietic system;
* Those who cannot cooperate with the treatment. Note: Those who meet any of the above items are not included in this trial.

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Week 4
  There are 19 sleep-related self-assessment questions that make up 7 components ranging from 0 to 3 points. The total score evaluation is: 0 to 5. Good sleep quality. 6 to 10. The sleep quality is okay. 11-15 Sleep quality is average; The sleep quality from 16 to 21 was very poor.
  The PSQI score reduction rate = (pre-treatment score - post-treatment score)/pre-treatment score ×100%. Cure: PSQI score reduction rate ≥75%. Effective rate: 50%≤ deduction rate < 75%. Effective: 25%≤ deduction rate < 50%. Invalid: PSQI deduction rate < 25%. The total effective rate = (number of cured patients + number of markedly effective patients + number of effective patients)/Total number of patients in this group of trials ×100%

SECONDARY OUTCOMES:
Traditional Chinese Medicine Syndrome Efficacy Assessment | Week 4
  According to the "Diagnostic and Therapeutic Criteria for Symptoms of Traditional Chinese Medicine", 11 observation indicators for insomnia of the heart andleen deficiency type were formulated. The TCM syndrome scoring table consists of 11 symptoms including sleep, dreaminess, palpitation, asthenia, dizziness,orexia, abdominal distension, loose stool, complexion, tongue image, and pulse condition. The first four items are scored according to 0, 2, 4 and 6 points, and the remaining seven items are scored according to 0-3 points, with a full score of 45 points. The higher the score, the consistent the symptoms are with the heart and spleen deficiency type.
Hamilton Anxiety Scale | Week 4
  The table includes 14 items, all of which adopt a 5-point scoring method of 0-4 points, 0 points: asymptomatic 1 point: mild; 2 points: moderate; 3 points: severe; 4 points: extremely severe.
Infrared thermal image acquisition | Week 4
  Compare the average temperature (℃) of the forehead and abdomen before and after treatment. A decrease in temperature after treatment indicates effectiveness. Through infrared thermal imaging, the sleep line on the forehead: ａ．Significantly effective: the sleep line completely disappears; ｂ．Effective: the sleep line changes from bilateral to unilateral;Ｃ．Ineffective: the sleep line does not change significantly. The total effective rate of sleep line improvement = (number of significantly effective cases number of effective cases) / number of cases × 100.0%.

IPD SHARING:
Plan to Share IPD: No